CLINICAL TRIAL: NCT05081232
Title: Radical Prostectomy (RAP): Prospective Trial Evaluating Return to Continence and Potency Following Radical Prostatectomy Using Novel Multi-Layer Perinatal Issue alloGraft
Brief Title: Continence and Potency Following Multi-Layer Perinatal Issue alloGraft
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will not be conducted
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00076844
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Recovery
Keywords: Multi-Layered Perinatal Tissue Allograft; Robot-Assisted Radical Prostatectomy; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: Male patients undergoing Robot-Assisted Radical Prostectomy and eligible will receive Human Umbilical Cord (UC) allograft. It is hypothesized that patients receiving UC allograft placed around the neurovascular bundle will facilitate earlier return to potency and continence compared to those that do not receive UC allografts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Umbilical Cord Allograft Recipients (Experimental): Male patients undergoing Robot Assisted Radical Prostectomy with bilateral nerve sparing technique will remain eligible to receive allograft during the surgery.
  Interventions: Device: MLG (Multi-Layered Perinatal Issue Allograft) Allograft

INTERVENTIONS:
Device: MLG (Multi-Layered Perinatal Issue Allograft) Allograft — MLG allografts contains more than 450 bioactive proteins including growth factors and cytokines known to modulate inflammation and promote tissue healing.
  MLG is supplied as sterile sheets having dimensions of 2cm x 2cm and a thickness of approximately 0.8-1.0mm thick.
  Participants receiving MLG will have it placed around the neurovascular bundle. Placement of the graft should not take over 5 minutes of time to impact overall surgical time length significantly.

SUMMARY:
The purpose of this research is to determine the effectiveness of using human Umbilical Cord (UC) allograft to help improve return to erectile function and bladder control in patients following robot-assisted radical prostatectomy (RARP).

DETAILED DESCRIPTION:
Participation in this study will involve MLG (Multi-Layered Perinatal Tissue Allograft) allograft, which is implanted during the surgery. This allograft is currently FDA approved and used for several type of surgeries.

The Multi-Layered Perinatal Tissue Allograft- (MLG) is processed from tissue according to the American Association of Tissue Banks (AATB) standards, and is regulated as a cell, tissue, or cellular or tissue-based product (HCT/P) under Section 361 of the Public Health Service Act. The grafts are distributed by Samaritan Biologics, LLC; an FDA-registered tissue bank.

The MLG allograft will be placed on each neurovascular bundle (NVB) bilaterally.

MLG is supplied as sterile sheets having dimensions of 2cm x 2cm and a thickness of approximately 0.8-1.0mm thick.

Participants receiving MLG will have it placed around the neurovascular bundle. Placement of the graft should not take over 5 minutes of time to impact overall surgical time length significantly.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects with at least age of 30 to 65
2. Primary diagnosis of prostate cancer selected for surgical intervention (Radical Prostatectomy)
3. Primary diagnosis of organ confined untreated prostate cancer
4. Planned elective radical prostatectomy with bilateral nerve sparing technique
5. Negative urinalysis within 30 days prior to date of surgery
6. Patient has no erectile dysfunction (SHIM Score < 14 ) prior to date of surgery
7. Patient has the willingness to comply with instruction of the investigator
8. Patient has the willingness to comply with follow-up surveys
9. Have ability to provide full written consent.

Exclusion Criteria:

1. High-risk cancer planned for neoadjuvant therapy, full or partial excision of neurovascular bundles
2. Is unable to comply with learning and documenting penile rehabilitation, including oral 5-phosphodiesterase inhibitor use, vacuum pump therapy use, and/or injectable medications
3. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study
4. Patients that have had prior hormonal therapy such as Lupron or oral anti-androgens
5. Patients with poor urinary control at baseline requiring the use of pads for leakage
6. Previous history of pelvic radiation
7. Previous history of simple prostatectomy or transurethral prostate surgery
8. Patients with obesity defined as BMI > 40 kg/m2
9. History of open pelvic surgery within 5 years except for hernia repair
10. Poorly controlled diabetes (A1C >8.5%)
11. Scheduled at the time of screening to undergo chemotherapy, radiation, hormone therapy, or open surgery during the study period
12. Any neurologic disorder or psychiatric disorder that might confound postsurgical assessments
13. Has any condition(s), which seriously compromises the subject's ability to participate in this study, sign consent, or has a known history of poor adherence with medical treatment
14. In the opinion of the PI, has a history of drug or alcohol abuse within last 12 months
15. Is allergic to Aminoglycoside antibiotics (such as Gentamicin and/or Streptomycin)
16. Received administration of an investigational drug within 30 days prior to study, and/or has planned administration of another investigational product or procedure during participation in this study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with Prostate Cancer
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Average time for return to potency | 1 month post-op
  Early recovery in potency will be measured as + 4 points of total Sexual Health Inventory for Men (SHIM) score in relation to baseline score. Return to potency will be defined as the ability to achieve an erection sufficient for intercourse more than 50% of the time or at least 50% rigidity post-robot-assisted radical prostatectomy (RARP) (Tool: SHIM, Q2 > 3)
Average time for return to potency | 3 month post-op
  Early recovery in potency will be measured as + 4 points of total SHIM score in relation to baseline score. Return to potency will be defined as the ability to achieve an erection sufficient for intercourse more than 50% of the time or at least 50% rigidity post-RARP (Tool: SHIM, Q2 > 3)
Average time for return to potency | 6 month post-op
  Early recovery in potency will be measured as + 4 points of total SHIM score in relation to baseline score. Return to potency will be defined as the ability to achieve an erection sufficient for intercourse more than 50% of the time or at least 50% rigidity post-RARP (Tool: SHIM, Q2 > 3)
Average time for return to potency | 12 month post-op
  Early recovery in potency will be measured as + 4 points of total SHIM score in relation to baseline score. Return to potency will be defined as the ability to achieve an erection sufficient for intercourse more than 50% of the time or at least 50% rigidity post-RARP (Tool: SHIM, Q2 > 3)
Average time for return to continence | 1-2 days post-op
  Return to continence will be defined as use of < 1 pad post-RARP
Average time for return to continence | 1 month post-op
  Return to continence will be defined as use of < 1 pad post-RARP
Average time for return to continence | 3 month post-op
  Return to continence will be defined as use of < 1 pad post-RARP
Average time for return to continence | 6 month post-op
  Return to continence will be defined as use of < 1 pad post-RARP
Average time for return to continence | 12 month post-op
  Return to continence will be defined as use of < 1 pad post-RARP

SECONDARY OUTCOMES:
Expanded prostate cancer index composite-26 (EPIC-26) Score | Months 1, 3, 6, and 12
  EPIC-26, contains five symptom domains (urinary incontinence, urinary irritative/obstructive, sexual, bowel, hormonal), scored from 0 (worst) to 100 (best)
Abdominal VAS (Visual Analog Scale) Pain Score | Post-op Days 1 and 2
  VAS score 0 -10: 0 indicating no abdominal pain to 10 as worst pain
Value analysis for a historical subset of patients who underwent same surgery as sexual health inventory for men (SHIM)-matched controls | Month 1 post-op
  Twenty-five patients who underwent bilateral nerve sparing in the past matched by preoperative SHIM to see how they did in comparison to study cohort will be measured as + 4 points of total SHIM score in relation to baseline score. Return to potency will be defined as the ability to achieve an erection sufficient for intercourse more than 50% of the time or at least 50% rigidity post-RARP (Tool: SHIM, Q2 > 3)
Costs of prescription | Month 12 post-op
  Oral Phosphodiesterase type 5 (PDE-5i), Intracavernosal injection, Alprostadil urethral suppository or future surgery (Inflatable penile prosthesis) to be recorded in the historical group of 25 patients. Overall expense will be measured by reviewing history. A market value of medication and treatment will be accounted. Post coverage out of pocket expense will not be reviewed separately.
Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) scores | Day 1 post-op
  Overall patient satisfaction Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) - composed of 29 items - the survey contains 19 core questions about critical aspects of patients' hospital experiences (communication with nurses and doctors, the responsiveness of hospital staff, the cleanliness and quietness of the hospital environment, communication about medicines, discharge information, overall rating of hospital, and would they recommend the hospital) - HCAHPS score is accounted as The "top-box" score indicates how often patients selected the most positive response category when asked about their hospital experience. The higher a hospital's "top-box" score, the higher it ranks.

CONTACTS AND LOCATIONS:
Overall Officials: Ram A Pathak, MD, Principal Investigator — Assistant Professor of Urology

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data from the study will be kept on password protected digital storage for at least three years following the project completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At least 3 years from study completion
Access Criteria: Contact the principal investigator (Dr. Ram Anil Pathak) or project manager (Sachin Nalin Vyas, MS,PhD)

REFERENCES:
- [Background] Neumaier MF, Segall CH Junior, Hisano M, Rocha FET, Arap S, Arap MA. Factors affecting urinary continence and sexual potency recovery after robotic-assisted radical prostatectomy. Int Braz J Urol. 2019 Jul-Aug;45(4):703-712. doi: 10.1590/S1677-5538.IBJU.2018.0704. PMID 31136108
- [Background] Carlsson S, Drevin L, Loeb S, Widmark A, Lissbrant IF, Robinson D, Johansson E, Stattin P, Fransson P. Population-based study of long-term functional outcomes after prostate cancer treatment. BJU Int. 2016 Jun;117(6B):E36-45. doi: 10.1111/bju.13179. Epub 2015 Jun 23. PMID 25959859
- [Background] Nelson CJ, Scardino PT, Eastham JA, Mulhall JP. Back to baseline: erectile function recovery after radical prostatectomy from the patients' perspective. J Sex Med. 2013 Jun;10(6):1636-43. doi: 10.1111/jsm.12135. Epub 2013 Apr 3. PMID 23551767
- [Background] Steineck G, Helgesen F, Adolfsson J, Dickman PW, Johansson JE, Norlen BJ, Holmberg L; Scandinavian Prostatic Cancer Group Study Number 4. Quality of life after radical prostatectomy or watchful waiting. N Engl J Med. 2002 Sep 12;347(11):790-6. doi: 10.1056/NEJMoa021483. PMID 12226149
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Castiglione F, Ralph DJ, Muneer A. Surgical Techniques for Managing Post-prostatectomy Erectile Dysfunction. Curr Urol Rep. 2017 Sep 30;18(11):90. doi: 10.1007/s11934-017-0735-2. PMID 28965315
- [Background] Menon M, Kaul S, Bhandari A, Shrivastava A, Tewari A, Hemal A. Potency following robotic radical prostatectomy: a questionnaire based analysis of outcomes after conventional nerve sparing and prostatic fascia sparing techniques. J Urol. 2005 Dec;174(6):2291-6, discussion 2296. doi: 10.1097/01.ju.0000181825.54480.eb. PMID 16280816
- [Background] Finley DS, Osann K, Skarecky D, Ahlering TE. Hypothermic nerve-sparing radical prostatectomy: rationale, feasibility, and effect on early continence. Urology. 2009 Apr;73(4):691-6. doi: 10.1016/j.urology.2008.09.085. Epub 2009 Feb 28. PMID 19250660
- [Background] Ogaya-Pinies G, Palayapalam-Ganapathi H, Rogers T, Hernandez-Cardona E, Rocco B, Coelho RF, Jenson C, Patel VR. Can dehydrated human amnion/chorion membrane accelerate the return to potency after a nerve-sparing robotic-assisted radical prostatectomy? Propensity score-matched analysis. J Robot Surg. 2018 Jun;12(2):235-243. doi: 10.1007/s11701-017-0719-8. Epub 2017 Jun 27. PMID 28656504
- [Background] Patel VR, Samavedi S, Bates AS, Kumar A, Coelho R, Rocco B, Palmer K. Dehydrated Human Amnion/Chorion Membrane Allograft Nerve Wrap Around the Prostatic Neurovascular Bundle Accelerates Early Return to Continence and Potency Following Robot-assisted Radical Prostatectomy: Propensity Score-matched Analysis. Eur Urol. 2015 Jun;67(6):977-980. doi: 10.1016/j.eururo.2015.01.012. Epub 2015 Jan 19. PMID 25613153
- [Background] Barski D, Gerullis H, Ecke T, Boros M, Brune J, Beutner U, Tsaur I, Ramon A, Otto T. Application of Dried Human Amnion Graft to Improve Post-Prostatectomy Incontinence and Potency: A Randomized Exploration Study Protocol. Adv Ther. 2020 Jan;37(1):592-602. doi: 10.1007/s12325-019-01158-3. Epub 2019 Nov 28. PMID 31782131
- [Background] Razdan S, Bajpai RR, Razdan S, Sanchez MA. A matched and controlled longitudinal cohort study of dehydrated human amniotic membrane allograft sheet used as a wraparound nerve bundles in robotic-assisted laparoscopic radical prostatectomy: a puissant adjunct for enhanced potency outcomes. J Robot Surg. 2019 Jun;13(3):475-481. doi: 10.1007/s11701-018-0873-7. Epub 2018 Sep 12. PMID 30209677
- [Background] Fetterolf DE, Snyder RJ. Scientific and clinical support for the use of dehydrated amniotic membrane in wound management. Wounds. 2012 Oct;24(10):299-307. PMID 25876055
- [Background] Koob TJ, Rennert R, Zabek N, Massee M, Lim JJ, Temenoff JS, Li WW, Gurtner G. Biological properties of dehydrated human amnion/chorion composite graft: implications for chronic wound healing. Int Wound J. 2013 Oct;10(5):493-500. doi: 10.1111/iwj.12140. Epub 2013 Aug 1. PMID 23902526
- [Background] Bullard JD, Lei J, Lim JJ, Massee M, Fallon AM, Koob TJ. Evaluation of dehydrated human umbilical cord biological properties for wound care and soft tissue healing. J Biomed Mater Res B Appl Biomater. 2019 May;107(4):1035-1046. doi: 10.1002/jbm.b.34196. Epub 2018 Sep 10. PMID 30199609